CLINICAL TRIAL: NCT06636175
Title: Early Phase I Evaluation of 64Cu-LLP2A for Imaging Hematologic Malignancies Part B
Brief Title: 64Cu-LLP2A for Imaging Hematologic Malignancies
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 202505198; R42CA257797 (NIH)
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma; Low-Grade Lymphoma; Follicular Lymphoma; Marginal Zone Lymphoma; Lymphoplasmacytic Lymphoma; Small Lymphocytic Lymphoma; Chronic Lymphocytic Leukemia
Keywords: PET; Imaging
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Intervention Model Description: For Cohort 1B, 6 healthy volunteers and 6 patients with either multiple myeloma (MM) or lymphoma will be recruited (healthy volunteers will be split equally with 3 men and 3 women enrolled, all efforts will be made to keep the number of subjects with MM and lymphoma enrolled equal to Cohort 1B but it will not be a requirement).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Pilot/Cohort 1B: Dosimetry 64Cu-LLP2A (Experimental): - Will be asked to undergo 64Cu-LLP2A-PET/CT imaging at up to three separate time points for purposes of calculating human dosimetry. Imaging time points will be dependent upon day of the week injection occurs:
  * Tuesday or Thursday injection: 0-60 minute multiple quick body scans + 120-180 min post injection body scan
  * Wednesday or Friday injection: 0-60 minute multiple quick body scans + 180-240 min post injection body scan
  * ALL PATIENTS: 15-28 hours post injection body scan on Wednesday (for Tuesday injection), Thursday (for Wednesday injection), Friday (for Thursday injection) or Saturday (for Friday injection)
  Interventions: Drug: 64Cu-LLP2A; Device: PET/CT
- Cohort 2B: Quantitative 64Cu-LLP2A (Experimental): - Will be asked to undergo dynamic PET/CT imaging centered over a known target lesion (as determined by other radiological imaging studies) beginning with 64Cu-LLP2A-PET/CT and continuing for a total of 60 minutes. An additional vertex to upper thigh body scan will be obtained between 60- and 180-minutes post injection or at the optimal imaging time point that was derived from cohort 1B.
  Interventions: Drug: 64Cu-LLP2A; Device: PET/CT

INTERVENTIONS:
Drug: 64Cu-LLP2A — 64Cu-LLP2A, will be manufactured following batch production record at the cyclotron GMP facility (Washington University School of Medicine GMP radiochemistry/cyclotron facility)
Device: PET/CT — The results of 64Cu-LLP2A-PET/CT will not be provided to the patient or the treating oncologist/surgeon unless, in the judgment of the principal investigator, the images demonstrate an unsuspected abnormality that may warrant further evaluation.

SUMMARY:
This phase of the protocol (protocol part B), seeks to evaluate the new formulation in healthy normal volunteers to confirm the new formulation provides comparable human dosimetry to which was seen and published in protocol part A. Additionally, the new formulation will be studied utilizing an expanded patient population to include patients with confirmed diagnosis of multiple myeloma (MM), low-grade lymphoma, or MM and lymphoma patients who are status post bone marrow transplant (BMT) with negative imaging and suspected recurrence.

ELIGIBILITY:
Inclusion Criteria Healthy Volunteer:

* Adult 18 years of age or older
* Able to give informed consent.
* Able to comprehend and willing to follow instructions for study procedures as called for by the protocol
* Capable of lying still and supine within the PET/CT scanner for up to 75 minutes.
* No illicit drug use or other inhaled drug use (including pharmacologic agents and illicit drugs) within the past year per self-reporting mechanisms.
* No history of claustrophobia or other condition that has previously or would interfere with completion of protocol specified imaging sessions.
* Not currently pregnant or nursing: Subject must be surgically sterile (has had a documented bilateral oophorectomy and/or documented hysterectomy), post-menopausal (cessation of menses for more than 1 year), non-lactating, or of childbearing potential for whom a urine pregnancy test (with the test performed within the 24 hour period immediately prior to administration of 64Cu-LLP2A) is negative.

Inclusion Criteria Hematological Malignancy:

* Clinical or pathologically defined MM or lymphoma including both newly diagnosed, relapsed or refractory disease:

  * Multiple Myeloma defined in accordance with the International Myeloma Working Group criteria
  * Low-grade lymphoma, including the following subtypes: follicular lymphoma, marginal zone lymphoma, lymphoplasmacytic lymphoma, small lymphocytic lymphoma/chronic lymphocytic leukemia
* Adult 18 years of age or older and able to provide informed consent
* Capable of lying still and supine within the PET/CT scanner for up to 75 minutes.
* No history of claustrophobia or other condition that has previously or would interfere with completion of protocol specified imaging sessions
* Not currently pregnant or nursing: Subject must be surgically sterile (has had a documented bilateral oophorectomy and/or documented hysterectomy), post-menopausal (cessation of menses for more than 1 year), non-lactating, or of childbearing potential for whom a urine pregnancy test (with the test performed within the 24 hour period immediately prior to administration of 64Cu-LLP2A) is negative
* Patients participating in imaging or therapeutic trials with investigational agents are eligible to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Organ dosimetry of participants | Through completion of PET/CT scans (estimated to be up to 2 days)
  Confirm organ dosimetry in healthy subjects and in patients with various hematological malignancies is consistent with prior formulation of 64Cu-LLP2A (all of Cohort 1 + up to 10 cohort 2 subjects). Average organ activity concentration will be measured, and decay corrected by utilizing regions of interest (ROIs) drawn around all organ visible on 64Cu-LLP2A images. Activity organ residence times will be calculated by numerical or analytical integration of the time-activity curves. Uptake/clearance functional fits of mono- or bi-exponential functions will be performed and analytical integration, accounted for physical decay, will be performed. The calculated residence times will be used with the program OLINDA/EXM for 64Cu and using the adult human (female and male) model to calculate the individual organ radiation dose, the whole-body dose and the effective dose.
Safety and tolerability of new formulation of 64Cu-LLP2A as measured by number of participants with adverse events | From beginning of administration of 64Cu-LLPA2A through last phone call assessment (up to 7 days total)
  Follow-up telephone call or in person visit to assess for self-reported adverse events associated with injection of 64Cu-LLP2A or PET/CT imaging. Additional chart review can be performed as needed.

SECONDARY OUTCOMES:
Evaluate the quality of PET images with new formulation 64Cu-LLP2A as measured by overall quality of PET images | Through completion of PET/CT scans (estimated to be up to 2 days)
  Overall, PET image quality will be graded visually (using 4-point scale with 1 being the worst and poor quality, not acceptable for diagnostic interpretation and 4 being good image quality, similar to routine clinical studies)
Evaluate the quality of PET images with new formulation 64Cu-LLP2A as measured by bone marrow uptake | Through completion of PET/CT scans (estimated to be up to 2 days)
  As measured by placing ROI and calculating SUVmax where SUVmax is a mathematical measurement of tumor burden seen on images and calculated by the following equation SUVmax= r / (a'/w) where r= radioactivity concentration in tumor (kBq/ml) as measured by the PET scanner within a defined region of interest, a'=the decay corrected amount of injected 64Cu-LLP2A and w= weight of the patient in grams
Evaluate the quality of PET images with new formulation 64Cu-LLP2A as measured by tumor/background ratio | Through completion of PET/CT scans (estimated to be up to 2 days)
  As measured by placing ROI and calculating SUVmax

CONTACTS AND LOCATIONS:
Overall Officials: Farrokh Dehdashti, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu